CLINICAL TRIAL: NCT03161561
Title: Mechanisms, Impact and Therapeutic Targeting of Bacterial Colonisation in COPD
Brief Title: Mechanisms and Impact of Bacterial Colonisation in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STH15949
Record Dates: First submitted 2017-05-11; First posted 2017-05-22 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Measurement of the capacity of primary phagocytes (neutrophils, monocytes and macrophages) isolated from COPD patients' blood or alveolar macrophages isolated from patients' lungs to carry out key host defence functions and compare these to similar cells isolated from age and sex-matched non-smokers or smokers without COPD as controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- capacity of primary phagocytes (Other): capacity of primary phagocytes isolated from COPD patients' blood to carry out key host defence functions and compare these to similar cells isolated from age and sex-matched non-smokers or smokers without COPD as controls.
  Interventions: Other: capacity of primary phagocytes

INTERVENTIONS:
Other: capacity of primary phagocytes — measurement of capacity of primary phagocytes (neutrophils, monocytes and macrophages) isolated from COPD patients' blood or alveolar macrophages isolated from patients' lungs to carry out key host defence functions and compare these to similar cells isolated from age and sex-matched non-smokers or smokers without COPD as controls.

SUMMARY:
COPD is a leading cause of lung disease and a common cause of hospitalisation, time off work and death. Smoking is the major factor associated with development of COPD. Nevertheless why some people develop COPD while others, including many smokers do not, is poorly understood. A central feature of COPD is accumulation of a particular type of white blood cell, the neutrophil, which is a key component in defence against bacterial infection in the lung airway. As disease progresses the small airways of many patients with COPD start to accumulate bacteria, which are normally lacking in the small airways of healthy individuals or smokers who lack COPD. The accumulation of bacteria in the smaller airways of many patients with COPD may be important to the development of the disease. Researchers will test if blood cells, which normally ingest and kill bacteria, have a reduced ability to perform this function in patients with COPD and whether the clearance of these blood cells after they have performed their role in protecting against infection is impaired. Researchers will relate these findings to the clinical features of COPD in a well-defined group of patients who have had extensive characterisation of their disease. In particular, researchers will relate this defect to the presence of frequent flares of disease, which lead to symptoms of wheezing and shortness of breath. Comparison will be made between blood cells obtained from the lung and from he blood to determine if the alterations are specific to the lung. Researchers will identify particular molecular alterations in the way these blood cells respond to bacteria and determine whether they can correct these alterations using agents, which are used to treat a range of different medical conditions, but which they predict might correct these alterations in function. The aim of this programme of work is ultimately to identify new ways in which to treat COPD and the agents, which the researchers demonstrate have the greatest potential to correct the abnormalities in cell function of patients with COPD, would in the future be studied in clinical trials.

DETAILED DESCRIPTION:
Work package one involves the consolidation and further characterisation of a number of pre-existing UK-based clinical cohorts of patients with COPD. This involves collection of epidemiological and physiological data from patients and controls to enable a complete definition of disease phenotype. Work package two will examine microbiological and innate immune parameters in this cohort to define whether innate immune defects underpin the susceptibility to infectious exacerbation and progression of airways disease. It will perform microbiological characterisation of each group and will look at the behaviour of groups who have frequent infectious exacerbations of disease as compared to those that do not. Work package three will measure lung injury and work package four will define physiological characteristics including chest wall muscle function in the cohort.

Our work will sit within work package two. Researchers will collect data from patients within the cohort and in patients whom they may recruit locally and add to the cohort. Researchers will also share samples with other work packages (academic and industry based collaborators) as required to enable correlation of our findings with other investigators in our work package or other work packages. This project, which sits within work-package two will measure the capacity of primary phagocytes (neutrophils, monocytes and macrophages) isolated from COPD patients' blood or alveolar macrophages isolated from patients' lungs to carry out key host defence functions and compare these to similar cells isolated from age and sex-matched non-smokers or smokers without COPD as controls.

ELIGIBILITY:
COPD Patients Inclusion Criteria:

aged 18-69 GOLD stage I or II have defined exacerbation frequency

Healthy Volunteers Inclusion Criteria:

age and sex matched to recruited COPD patients either non-smokers or smokers with at least 10 years history of smoking at least 10 cigarettes per day.

COPD Patients Exclusion Criteria:

Individuals known to have active malignancy, immunosuppression, diabetes mellitus, chronic kidney disease or hepatic failure.

Individuals with a history of anaemia Individuals who have donated >200 ml of blood for any reason within the last 6months Individuals who are pregnant or breast feeding. Current participation in any other clinical trial, except those directly relating to this cohort and study.

Inability to communicate in English or convey willingness to participate.

For bronchoscopy - any active lung condition including:

Any active acute lung infection (with the exception of asymptomatic pulmonary colonisation) or malignancy Significant coexisting interstitial lung disease or additional pulmonary diagnosis in addition to COPD Significant interstitial lung disease (on radiological and PFT criteria) Any significant abnormality on CXR that would contraindicate bronchoscopy

Healthy Volunteers Exclusion Criteria:

Individuals who have had a febrile illness or other symptoms of acute infectious illness (respiratory, enteric or soft tissue) within the last 2 weeks.

Chronic or acute respiratory disease. Any chronic medical condition or receipt of regular prescription medication other than the oral contraceptive pill.

Individuals who have received a vaccine in the past two weeks. Individuals with a history of anaemia or any symptoms (shortness of breath, chronic fatigue, chest pain or pallor) suggestive of possible anaemia or haemoglobin below the lower limit of sex adjusted normal range.

Individuals who have donated >200 ml of blood for any reason within the last 6 months.

Individuals who are pregnant or breast feeding. Current participation in any clinical trial. Inability to communicate in English or convey willingness to participate

For bronchoscopy - any active lung condition including:

Any lung infection Asthma

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-11-16 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
JC-1 assay of phagocytosis | day 0
  Using preliminary data derived from the performance of one of the assays to be performed to measure apoptosis on these patient's macrophages, the JC-1 assay of loss of inner mitochondrial transmembrane potential

CONTACTS AND LOCATIONS:
Overall Officials: Paul Collini, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No